CLINICAL TRIAL: NCT00104260
Title: A Phase 2, Multicenter, Open-Label Study to Evaluate the Response to and Safety of an 8-Day Course of Phenoptin™ Treatment in Subjects With Phenylketonuria Who Have Elevated Phenylalanine Levels
Brief Title: Study to Evaluate the Response to and Safety of an 8-Day Course of Phenoptin™ Treatment in Subjects With Phenylketonuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-001
Record Dates: First submitted 2005-02-24; First posted 2005-02-25 (Estimated); Last update posted 2007-04-09 (Estimated); Status verified 2007-04

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

INTERVENTIONS:
Drug: sapropterin dihydrochloride

SUMMARY:
The primary objective is to evaluate the degree and frequency of response to Phenoptin™ (sapropterin dihydrochloride), as demonstrated by a reduction in blood phenylalanine (Phe) level among subjects with phenylketonuria (PKU) who have elevated Phe levels. A secondary objective of this study is to evaluate the safety of Phenoptin™ treatment in this subject population, and identify individuals in this subject population who respond to Phenoptin™ treatment with a reduction in blood Phe level.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 8 years
* Blood Phe level >/= 450 umol/L at screening
* Clinical diagnosis of PKU with hyperphenylalaninemia documented by past medical history of at least one blood Phe measurement >/= 360 umol/L (6 mg/dL)
* Willing and able to provide written informed consent or, in the case of subjects under the age of 18, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained
* Negative urine pregnancy test at screening (non-sterile females of child-bearing potential only)
* Male and Female subjects of childbearing potential childbearing potential (if sexually active and non-sterile) must be using acceptable birth control measures, as determined by the investigator, and willing to continue to use acceptable birth control measures while participating in the study
* Willing and able to comply with study procedures
* Willing to continue current diet unchanged while participating in the study

Exclusion Criteria:

* Perceived to be unreliable or unavailable for study participation or, if under the age of 18, have parents or legal guardians who are perceived to be unreliable or unavailable
* Use of any investigational agent within 30 days prior to screening, or requirement for any investigational agent or vaccine prior to completion of all scheduled study assessments
* Pregnant or breastfeeding, or considering pregnancy
* ALT > 5 times the upper limit of normal (i.e., Grade 3 or higher based on World Health Organization Toxicity Criteria) at screening
* Concurrent disease or condition that would interfere with study participation or safety (e.g., seizure disorder, oral steroid-dependent asthma or other condition requiring oral or parenteral corticosteroid administration, or insulin-dependent diabetes, or organ transplantation)
* Serious neuropsychiatric illness (e.g., major depression) not currently under medical control
* Requirement for concomitant treatment with any drug known to inhibit folate synthesis (e.g., methotrexate)
* Concurrent use of levodopa
* Clinical diagnosis of primary BH4 deficiency

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700
Dates: Start 2004-12; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the degree and frequency of response to Phenoptin™, as demonstrated by a reduction in blood Phe level among subjects with PKU who have elevated Phe levels

SECONDARY OUTCOMES:
Evaluate the safety of Phenoptin™ treatment in this subject population, and identify individuals in this subject population who respond to Phenoptin™ treatment with a reduction in blood Phe level

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Los Angeles, California
  - Oakland, California
  - New Haven, Connecticut
  - Chicago, Illinois
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Salt Lake City, Utah
  - Madison, Wisconsin